CLINICAL TRIAL: NCT03572465
Title: Quantitative Ultrasound Techniques for Diagnosis of Nonalcoholic Steatohepatitis
Acronym: QUS in NASH
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: CE 18.109
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD); Nonalcoholic Steatohepatitis (NASH)
Keywords: Chronic liver disease; Fibrosis; Elastography; Ultrasound; Magnetic resonance elastography; Diagnostic performance; Sensitivity and specificity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Hypersensitivity | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Liver biopsy specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NAFLD, NASH patients: All patients enrolled will undergo:
  * Acoustic Radiation Force Impulse (ARFI)
  * Magnetic Resonance Elastography (MRE)
  Interventions: Device: Acoustic radiation force impulse (ARFI), magnetic resonance elastography (MRE)
- Non-obese volunteers: All patients enrolled will undergo:
  * Acoustic Radiation Force Impulse (ARFI)
  * Magnetic Resonance Elastography (MRE)
  Interventions: Device: Acoustic radiation force impulse (ARFI), magnetic resonance elastography (MRE)

INTERVENTIONS:
Device: Acoustic radiation force impulse (ARFI), magnetic resonance elastography (MRE) — Acoustic Radiation Force Impulse (ARFI), Magnetic Resonance Elastography (MRE)

SUMMARY:
Nonalcoholic fatty liver disease is the most common liver disease in Western countries, due in large part to its association with type 2 diabetes and obesity. The more advanced form of this disease is known as nonalcoholic steatohepatitis (NASH). If left untreated, NASH can evolve to cirrhosis, the late stage of fibrosis. Once cirrhosis is established, patients are at increased risk of developing gastrointestinal bleeding, liver cancer and liver failure that may require transplantation. A liver biopsy is currently needed to diagnose the severity of fatty liver disease but this is usually not indicated in asymptomatic patients. This procedure requires the insertion of a needle inside the liver to remove a small piece of tissue for examination under microscope. Liver biopsy is an invasive procedure with a small risk of major complications such as bleeding in 0.5% of cases. It is also affected by sub-optimal sampling leading to diagnostic errors

Ultrasound is optimum for screening patients with or without symptoms because it is a safe and widely available technology to scan the whole liver. Members of our team have developed Advanced ultrasound techniques that provide unique information not possible with state-of-the-art techniques. Unlike liver biopsy, these techniques would be applicable even in asymptomatic patients because it is non-invasive. This research proposal proposes a novel approach for diagnosis of NASH and will be the first study to measure individual components of NASH (fat, inflammation and fibrosis) with quantitative ultrasound (QUS) scores. This study is timely because NASH is the second leading cause of liver transplantation in North America and is predicted to become the leading indication in the near future.

DETAILED DESCRIPTION:
BACKGROUND - Nonalcoholic fatty liver disease (NAFLD) is the most prevalent liver disease in Western countries. The more advanced form, nonalcoholic steatohepatitis (NASH) may evolve to fibrosis, cirrhosis, liver failure and liver cancer. Liver biopsy is the current reference standard for diagnosis of NASH. However, its invasiveness prevent its use for large-scale screening and diagnosis. Members of our team have developed innovative quantitative ultrasound (QUS) techniques (shear wave viscoelastography and sub-resolution cellular imaging) that have a high diagnostic potential. Advantages over magnetic resonance (MR) include the ability to characterize viscosity, cellular organizations and cost-effectiveness. We hypothesize that a combination of QUS techniques offering complementary assessment of tissue characteristics will differentiate NASH from NAFLD and quantify evolving grades of liver fat, inflammation and fibrosis.

OBJECTIVES - Primary objective: 1) Determine the accuracy of QUS parameters for diagnosis of NASH. Secondary objectives: 2) Determine the diagnostic accuracy of QUS for grading histology-determined liver fat, inflammation and fibrosis. 3) Compare the diagnostic accuracy of QUS and MR techniques for liver fat quantification.

Hypotheses: We hypothesize that QUS methods, including viscoelasticity, homodyned-K parameters and attenuation parameters can characterize properties of tissues encountered in NASH (including liver fat, inflammation and fibrosis).

METHODOLOGY - Design: This will be a cross-sectional imaging trial to evaluate the diagnostic accuracy of QUS techniques in 10 non-obese volunteers and 92 patients, using histopathology as the reference standard for patients. Paired index tests QUS-based (mechanical and cellular parameters) and MR-based (mechanical parameters and relaxation times reflecting tissue content) techniques will be performed as research procedures in close temporal proximity to the reference test (liver biopsy).

Inclusion criteria: Consecutive adult patients with known or suspected NAFLD or NASH undergoing a liver biopsy for clinical indications.

Exclusion criteria: Contraindication to MR, refusal to participate, any other cause of chronic liver disease or prior liver transplantation.

Data analysis: Random forest classifier to develop a predictive model. Cross-validated receiver operating characteristic curve analysis, sensitivity and specificity to assess diagnostic accuracy.

RATIONALE AND IMPACT - NASH has become the second leading cause of liver transplantation in North America and is predicted to become the leading indication in the near future. While liver biopsy is the established reference standard for NASH diagnosis and MR constitutes a noninvasive alternative, they are both impractical for large-scale application. Thus, there is an urgent need to investigate non-invasive and cost-effective techniques for diagnosis of NASH. Our proposed QUS techniques are experimental and currently not available on clinical US systems. A major impact of this work, for patients and medical institutions, will be to lower the need for liver biopsy, the risk of complications and reduce the cost for NASH diagnosis while providing quantitative therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old at screening;
* Able to comprehend and willingness to provide voluntary consent;
* Understand French or English;
* NAFLD/NASH subjects:

  * Have a suspected or known NAFLD or NASH;
  * Must undergo a liver biopsy as part of their clinical standard of care
* Non-NAFLD volunteers:

  * Do not have a suspected or known NAFLD or NASH

Exclusion Criteria:

* Are pregnant or trying to become pregnant;
* Have a weight or girth preventing them from entering the MR magnet bore;
* Are unable to understand or unwilling to provide written informed consent for this study;
* Non-NAFLD volunteers:

  * Have risk factors for developing liver steatosis (type 2 diabetes mellitus, alcohol consumption >60g of alcohol per day, lipogenic medication and body mass index >25 kg/m2);
  * Have a liver steatosis (defined as MRI-proton density fat fraction <5%);
* NAFLD/NASH subjects:

  * Have other causes of chronic liver disease;
  * Have a liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is adults with NAFLD or NASH and healthy volunteers (non-NAFLD subjects). For the purpose of this study, we will recruit NAFLD or NASH patients seen at the hepatology clinic of CHUM, a tertiary care center, and from the McGill University Health Centre (MUHC). Non-NAFLD volunteers will be recruited at the CHUM among the personnel.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Fibrosis stage | Within 6 weeks of liver biopsy
  Measure of fibrosis stage using histology

SECONDARY OUTCOMES:
Liver stiffness determined by ARFI | Within 6 weeks of liver biopsy
  Measure of liver stiffness using Acoustic Radiation Force Impulse (ARFI)-determined liver stiffness
Liver stiffness determined by MRE | Within 6 weeks of liver biopsy
  Measure agnetic Resonance Elastography (MRE)-determined
Magnetic Resonance Imaging (MRI)-based Proton Density Fat Fraction (PDFF) | Within 6 weeks of liver biopsy
Staging liver fibrosis | Within 6 weeks of liver biopsy
  Measure of staging liver fibrosis using magnetic Resonance Imaging (MRI) cine-tagging of cardiac-induced motion

CONTACTS AND LOCATIONS:
Overall Officials: An Tang, MD, MSc, Study Director — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada